CLINICAL TRIAL: NCT02538185
Title: Intradermal Rabies Immunization Using NanoJect: A Comparative Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Giuseppe Pantaleo, Prof. G. Pantaleo, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VIC-NANO-001
Record Dates: First submitted 2015-07-08; First posted 2015-09-02 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Intradermal (ID) Vaccination Device
MeSH Terms: interventions — Needles

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vaccine injected ID with classical syringe (Placebo Comparator): Right forearm, ID with NanoJect device (DebioJect™) filled with placebo (0.1mL);
  Left forearm, ID with classical syringe filled with vaccine (0.1mL);
  Non-dominant deltoid, Intramuscular (IM) with classical syringe filled with placebo (0.5mL).
  Interventions: Device: NanoJect device (DebioJect™); Device: Classical syringe (1mL Becton Dickinson (BD) Luer-Lock™) with a 25 Guage (G) needle (Terumo® Neolus); Device: Classical syringe (1mL BD Luer-Lock™) with a 22G needle (Terumo® Neolus); Drug: Vaccin rabique Pasteur®; Drug: Placebo
- Vaccine injected ID with NanoJect device (DebioJect™) (Active Comparator): Right forearm, ID with NanoJect device (DebioJect™) filled with vaccine (0.1mL);
  Left forearm, ID with classical syringe filled with placebo (0.1mL);
  Non-dominant deltoid, IM with classical syringe filled with placebo (0.5mL).
  Interventions: Device: NanoJect device (DebioJect™); Device: Classical syringe (1mL Becton Dickinson (BD) Luer-Lock™) with a 25 Guage (G) needle (Terumo® Neolus); Device: Classical syringe (1mL BD Luer-Lock™) with a 22G needle (Terumo® Neolus); Drug: Vaccin rabique Pasteur®; Drug: Placebo
- Vaccine injected IM with classical syringe (Placebo Comparator): Right forearm, ID with NanoJect device (DebioJect™) filled with placebo (0.1mL);
  Left forearm, ID with classical syringe filled with placebo (0.1mL);
  Non-dominant deltoid, IM with classical syringe filled with vaccine (0.5mL).
  Interventions: Device: NanoJect device (DebioJect™); Device: Classical syringe (1mL Becton Dickinson (BD) Luer-Lock™) with a 25 Guage (G) needle (Terumo® Neolus); Device: Classical syringe (1mL BD Luer-Lock™) with a 22G needle (Terumo® Neolus); Drug: Vaccin rabique Pasteur®; Drug: Placebo

INTERVENTIONS:
Device: NanoJect device (DebioJect™) — The investigational device used in this study is the NanoJect™ device developed by Debiotech company.
Device: Classical syringe (1mL Becton Dickinson (BD) Luer-Lock™) with a 25 Guage (G) needle (Terumo® Neolus) — The comparator device used for standard ID injections is a classical syringe (1mL BD Luer-Lock™) with a 25G needle (Terumo® Neolus)
Device: Classical syringe (1mL BD Luer-Lock™) with a 22G needle (Terumo® Neolus) — The comparator device used for standard IM injections is a classical syringe (1mL BD Luer-Lock™) with a 22G needle (Terumo® Neolus)
Drug: Vaccin rabique Pasteur®
Drug: Placebo — Sodium Chloride (NaCl) 0,9%; B. Braun

SUMMARY:
The study is planned as a single-center, randomized, double-blind placebo-controlled, comparative Phase I, first-in-man study to assess the safety and tolerability of the NanoJect™ device, and the immunogenicity of the rabies vaccine "Vaccin rabique Pasteur®" delivered with the NanoJect™ device by ID route.

DETAILED DESCRIPTION:
This study will enroll 66 volunteers randomly assigned to one of the three study arms. Each volunteer will receive three injections at each of three vaccination visits. Total study duration per volunteer is 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Has completed the written informed consent process.
* Is male or female aged 18 years and 50 years.
* Agrees to stay in contact with the study site for the duration of the study, provide updated contact information as necessary, and has no current plans to move from the study area for the duration of the study.
* Agrees to avoid elective surgery for the duration of the study.
* For female subjects: agrees to avoid pregnancy through the duration of the study.
* Is in good general health, confirmed by medical history, physical examination and screening laboratory tests.

Exclusion Criteria:

* Oral body temperature 37.5 Celcius (C).
* History or evidence of rabies vaccination or rabies contact.
* Abnormal CBC (Complete Blood Count) laboratory values (>10% above Upper Limit of Normal (ULN) or >10% below Lower Limit of Normal (LLN)) and abnormal biochemistry values from blood collected at screening (>10% above ULN or >10% below LLN). Analysis can be repeated upon request of the clinician.
* History or evidence of autoimmune disease.
* History or evidence of any past, present, or future possible immunodeficiency state, including HIV 1 infection.
* History or evidence of chronic hepatitis, including presence of anti-hepatitis B core antibodies or anti-hepatitis C antibodies.Participation in any other investigational study during the study period.
* Received immunoglobulin or blood products within 90 days prior to study visit 2.
* Received any investigational drug therapy or investigational vaccine within 180 days prior to study.
* Received any licensed vaccine within 45 days prior to study visit 2 (note: the use of licensed vaccines medically indicated during the study is permitted at any time).
* History or evidence of any treatment that, in the opinion of the investigator, may interfere with the vaccine response or compromise the safety of the subject.
* Received Chloroquin and/or Proguanil treatment within 420 days prior to study.
* Use of immunosuppressive drugs or anticoagulants.
* All female subjects: currently pregnant or lactating/nursing; positive screening urine pregnancy test; or positive urine pregnancy test on the day of any study vaccination
* History or evidence of allergic disease or reaction that, in the opinion of the investigator, may compromise the safety of the subject (Notably: allergy to active principle, excipients, polymyxin B, Streptomycin, Neomycin).
* History or evidence of dermatologic disease that, in the opinion of the investigator, may interfere with the assessment of injection site reactions.
* History or evidence of any other acute or chronic disease that, in the opinion of the investigator, may interfere with the evaluation of the safety or immunogenicity of the vaccine or compromise the safety of the subject.
* Medical, psychiatric, occupational, or substance abuse problems that, in the opinion of the investigator, will make it unlikely that the subject will comply with the protocol.
* History or evidence of any brain disease that, in the opinion of the investigator, may interfere with the vaccine and compromise the safety of the subject.
* Abnormal urinalysis at the screening visit that, in the opinion of the investigator, is clinically significant.
* Skin coloration (skin color, tattoo, freckles) that, in the opinion of the investigator, could interfere with injection reactogenicity assessment.
* Body Mass Index (BMI)<= 18 and => 33 (weight/height2). Immediate need of rabies immunization.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2013-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events as a Measure of Safety and Tolerability | At the end of the study, at Day 56 (visit 5).
Pain Scores at needle insertion and at product injection as measured by the Visual Analog Scale | At each product injection: Day 0 (visit 2), Day 7 (visit 3) and at Day 28 (visit 4).
Pain following product injection as a Measure of Safety and Tolerability | Change between baseline and 30 minutes after each injection, the evening after each injection and daily up to 3 days after each injection (product injection visits: Day 0 (visit 2), Day 7 (visit 3) and at Day 28 (visit 4)).
Redness following product injection as a Measure of Safety and Tolerability | Change between baseline and 30 minutes after each injection, the evening after each injection and daily up to 3 days after each injection (product injection visits: Day 0 (visit 2), Day 7 (visit 3) and at Day 28 (visit 4)).
Pruritus following product injection as a Measure of Safety and Tolerability | Change between baseline and 30 minutes after each injection, the evening after each injection and daily up to 3 days after each injection (product injection visits: Day 0 (visit 2), Day 7 (visit 3) and at Day 28 (visit 4)).

SECONDARY OUTCOMES:
Titers of Immunoglobulin G (IgG) anti-rabies antibodies analyzed by Rapid Fluorescent Focus Inhibition Test (RFFIT) as a measure of Immunogenicity | Change between baseline and last study visit: Day 56 (visit 5).

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Pantaleo, Principal Investigator — CHUV